CLINICAL TRIAL: NCT06577805
Title: A Retrospective Cohort Study of Prospectively Collect the Outcomes of Recipients After Robot-assisted Kidney Transplantation
Brief Title: The Outcomes of Living Donor Robotic Assisted Kidney Transplantation
Acronym: RAKT
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Tao Lin, Professor Tao Lin, West China Hospital
Other Study IDs: WestChina-RAKT
Record Dates: First submitted 2024-08-24; First posted 2024-08-29 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Kidney Transplant; Complications; Renal Failure Chronic
Keywords: robotic surgery
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- grafts with a single artery (GSA): recipients of grafts with a single artery undergoing living donor robotic-assisted kidney transplantation
- grafts with multiple single arteries (GMA): recipients of grafts with multiple renal arteries undergoing living donor robotic-assisted kidney transplantation

SUMMARY:
The technology for robot-assisted kidney transplantation (RAKT) has become increasingly advanced, with numerous studies demonstrating comparable outcomes between RAKT surgery and open surgery. This advancement is particularly noteworthy as it extends its suitability to transplant patients with obesity. It will be important to explore the results of robot-assisted kidney transplantation as compared with open surgery or within cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. living-donor kidney transplant recipients
2. receiving standard triad immunosuppressive regimen

Exclusion Criteria:

1. active infection
2. multi-organ transplantation
3. malignancy history in the donor and recipient
4. human immunodeficiency virus infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage 5 chronic kidney disease undergoing living robot-assisted kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The graft function of recipients | in the follow-up period，about six months to one year
  the graft function of recipients per month after transplant surgery, assessed by the serum creatinine (umol/L) and estimated glomerular function rate (eGFR).

SECONDARY OUTCOMES:
total operative time | about 150 minutes to 300 minutes
  The time from the beginning of the procedure to the end of the procedure (minute)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang Y, Zhang H, Yin S, Li Y, Zeng J, Lin T, Song T. The Early Outcomes of Robotic-Assisted Kidney Transplantation Using Grafts With Multiple Arteries From a High-Volume Center: A Retrospective Cohort Study. Clin Transplant. 2025 Oct;39(10):e70328. doi: 10.1111/ctr.70328. PMID 40988626